CLINICAL TRIAL: NCT06108804
Title: Comparative Effects of Mulligan Pain Release Phenomenon With and Without Tapping in Management of Patellofemoral Pain Syndrome
Brief Title: Comparative Effects of Mulligan Pain Release Phenomenon With and Without Tapping in Patellofemoral Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0142
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; mulligan's pain release phenomenon; tapping; kujala scale
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: A parallel study is a type of clinical study in which two or more groups of participants receive different interventions.
Who Masked: Participant
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mulligan pain release phenomenon with tapping. (Experimental): Participants in group A will receive mulligan pain release phenomenon with tapping.
  Interventions: Other: mulligan pain release phenomenon with tapping
- mulligan pain release phenomenon (Active Comparator): Participants in group B will receive mulligan pain release phenomenon
  Interventions: Other: mulligan pain release phenomenon

INTERVENTIONS:
Other: mulligan pain release phenomenon with tapping — Participants in Group A will receive mulligan pain release phenomenon with tapping.First, demographic information will be gathered, pain severity will be measured using NPRS, knee joint range of motion (flexion/extension) will be measured using a goniometer, and functional limitation will be evaluated using a Kujala score.Two sessions of treatment per week with a total of eight session will be given in four weeks
  Other Names: tapping
  Arms: mulligan pain release phenomenon with tapping.
Other: mulligan pain release phenomenon — Two sessions of treatment per week with a total of eight session will be given in four weeks.Group B will receive mulligan pain release phenomenon only. First, demographic information will be gathered, pain severity will be measured using NPRS. knee joint range of motion (flexion/extension) will be measured using a goniometer, and functional limitation will be evaluated using a Kujala score.
  Arms: mulligan pain release phenomenon

SUMMARY:
The aim of this study is to compare the effects of mulligan pain release phenomenon with or without Tapping in management of Patellofemoral pain syndrome

DETAILED DESCRIPTION:
Patellofemoral pain syndrome is a general phrase that refers to discomfort in the Patellofemoral joint and associated soft tissues, including the kneecap, tendons, and ligaments.

In 2019, a comparative study conducted. They pick 30 respondents randomly, who met the study's inclusion requirements and expressed a willingness to participate. They were split into two groups; fifteen subjects per group. Each group received treatment for four weeks, with sessions occurring every other day. PRP with Kinesiotaping is in Group A(n=15), and traditional therapy is in Group B(n=15). Both groups underwent ultrasonic treatment and VMO strengthening. Data analysis was carried out statistically using paired t tests within groups and unpaired t tests across groups. The study's findings indicated that both groups of therapy were successful, however PRP combined with Kinesiotaping significantly reduced pain and improved functional limits in patients with persistent Patellofemoral OA.

In 2020, a double blind RCT study conductred. Based on the mechanical correction approaches, 43 women with at least a 3-month history of PFPS were randomized into three groups: KT for patellar medialization, KT for lateral rotation of the femur and tibia, and the control group. The identical 12-week muscle- building and motor-control exercises were administered to all groups. The numerical pain rating scale (NPRS) at rest and during exertion, the kujala score (AKPS), and the single jump hop test were used to assess knee pain and function at baseline, at 6 weeks, at the end of therapy (12 weeks), and during the 12-week follow-up. Results of the study showed that, in the 6-week and 12-week follow-ups, there were clinically significant differences between the KT with lateral rotation of femur and tibia and the control group in terms of the AKPS and NPRS scores during effort. Pain and function significantly improved in all groups (within group).

Patellofemoral pain syndrome is a prevalent issue among the adults due to prolong sitting, ascending or descending stairs frequently, crouching and walking. The majority of research studies have primarily focused on other age groups, such as older adults or adolescents and very little study was done regarding this issue among young adults. To the best of our knowledge although in the past many studies have worked on mulligan pain release phenomenon with mobilization, or exercise therapy have been practiced in the treatment of Patellofemoral pain syndrome were found effective individually, but there is a lack of comprehensive studies including randomized clinical trials directly comparing the mulligan pain release phenomenon with or without taping on management of Patellofemoral pain syndrome. This RCT will aims to evaluate the effectiveness of two commonly utilized techniques, Mulligan pain release phenomenon and taping will ascertain that if two of these, Mulligan pain release phenomenon and taping, may have different effects on the Patellofemoral pain syndrome, knee range of motion and pain in young population with PFPS.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 40 years
* Both male and female
* NPRS>3
* AKPS ≥6
* ROM<135 ° rarely. Knee range of motion is usually normal in patients of Patellofemoral pain syndrome.
* Positive patellar grind test
* Adults having anterior knee pain from previous duration of 2-3 months which is aggravated by walking, stairs ambulation or prolong sitting.

Exclusion Criteria:

* Recent fracture/trauma
* Acute diseased condition
* Knee surgery
* Tumor or infection around the knee
* Rheumatoid Arthritis
* Pregnancy
* Any malformation or joint hypermobility
* patellar tendon pathology

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4th week
  Changes from baseline. The NPRS is a self-reporting or clinician-administered measuring tool that has extreme values ranging from "no pain" to "severe pain", on either horizontal or vertical line of scale.NPRS which is an eleven point scale in which no pain (score 0) and highest pain (score 10)
Knee Flexion Range of Motion | 4th week
  Changes from baseline. The measurement of joint range of motion (ROM) is an essential procedure used in physical therapy, known as goniometry
Knee Extension Range of Motion | 4th week
  Changes from baseline. The measurement of joint range of motion (ROM) is an essential procedure used in physical therapy, known as goniometry
Kujala Score (AKPS) | 4th week
  Changes from baseline. Kujala score is a 13 items, self-report questionnaire for the patients having Patellofemoral pain syndrome (PFPS). Kujala has been demonstrated to be valid and reliable in PFPS patients and can be utilized for clinical evaluation as well as research work.

CONTACTS AND LOCATIONS:
Overall Officials: Humera Mubashar, MS, Principal Investigator — Riphah International University
Locations (1):
- Kot Khawaja Saeed Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang WD, Chen FC, Lee CL, Lin HY, Lai PT. Effects of Kinesio Taping versus McConnell Taping for Patellofemoral Pain Syndrome: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2015;2015:471208. doi: 10.1155/2015/471208. Epub 2015 Jun 21. PMID 26185517
- [Background] Baldon Rde M, Nakagawa TH, Muniz TB, Amorim CF, Maciel CD, Serrao FV. Eccentric hip muscle function in females with and without patellofemoral pain syndrome. J Athl Train. 2009 Sep-Oct;44(5):490-6. doi: 10.4085/1062-6050-44.5.490. PMID 19771287
- [Background] Taunton JE, Ryan MB, Clement DB, McKenzie DC, Lloyd-Smith DR, Zumbo BD. A retrospective case-control analysis of 2002 running injuries. Br J Sports Med. 2002 Apr;36(2):95-101. doi: 10.1136/bjsm.36.2.95. PMID 11916889
- [Background] Pal S, Draper CE, Fredericson M, Gold GE, Delp SL, Beaupre GS, Besier TF. Patellar maltracking correlates with vastus medialis activation delay in patellofemoral pain patients. Am J Sports Med. 2011 Mar;39(3):590-8. doi: 10.1177/0363546510384233. Epub 2010 Nov 12. PMID 21076015
- [Background] Leibbrandt DC, Louw QA. The use of McConnell taping to correct abnormal biomechanics and muscle activation patterns in subjects with anterior knee pain: a systematic review. J Phys Ther Sci. 2015 Jul;27(7):2395-404. doi: 10.1589/jpts.27.2395. Epub 2015 Jul 22. PMID 26311990
- [Background] Logan CA, Bhashyam AR, Tisosky AJ, Haber DB, Jorgensen A, Roy A, Provencher MT. Systematic Review of the Effect of Taping Techniques on Patellofemoral Pain Syndrome. Sports Health. 2017 Sep/Oct;9(5):456-461. doi: 10.1177/1941738117710938. Epub 2017 Jun 15. PMID 28617653
- [Background] Arrebola LS, Teixeira de Carvalho R, Lam Wun PY, Rizzi de Oliveira P, Firmo Dos Santos J, Coutinho de Oliveira VG, Pinfildi CE. Investigation of different application techniques for Kinesio Taping(R) with an accompanying exercise protocol for improvement of pain and functionality in patients with patellofemoral pain syndrome: A pilot study. J Bodyw Mov Ther. 2020 Jan;24(1):47-55. doi: 10.1016/j.jbmt.2019.05.022. Epub 2019 May 22. PMID 31987562